CLINICAL TRIAL: NCT01719367
Title: Genetically Determined Response to Atenolol in Patients With Persistent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130298
Record Dates: First submitted 2012-10-29; First posted 2012-11-01 (Estimated); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Atrial Fibrillation
Keywords: Baseline (pre-atenolol); Post-atenolol
MeSH Terms: conditions — Atrial Fibrillation | interventions — Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Atenolol (Experimental): Patients will undergo a standardized, graded exercise protocol before and after receiving a dose of oral atenolol.
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Atenolol

SUMMARY:
Atrial fibrillation (AF), the most common sustained heart rhythm disorder, is becoming increasingly prevalent in the Western world. The number of people with AF in the United States is projected to roughly double by the year 2050, to an estimated 6-12 million. For many patients with AF, rate control with atrioventricular (AV) node blockers is a widely accepted therapeutic strategy. These agents control heart rate, thus preventing symptoms and systolic heart failure associated with tachycardia due to a rapid ventricular response to AF. Beta-blockers are widely accepted as first line agents for rate control in AF, especially when patients have concomitant hypertension (HTN), coronary artery disease, cardiomyopathies, or heart failure (HF). As a class, beta-blockers are among the most commonly prescribed cardiovascular medications.

Among patients with AF treated with beta-blockers, the heart rate (HR) response varies substantially. Sometimes, adequate rate control can be achieved by titration of the beta-blocker dose; but frequently, additional AV nodal blockers and/or digoxin are necessary. In some cases, adequate rate control cannot be achieved even with the simultaneous use of multiple AV nodal blockers, necessitating mechanical ablation of the AV node and permanent pacemaker implantation.

Patient-specific variables that influence the response to beta-blockers include comorbid conditions, weight, age, and level of physical activity. Ethnic differences in the response to beta-blockers for the treatment of HTN and HF are well-described. However, the contribution of genetic variants to beta-blocker efficacy in AF is unknown. We propose to study whether the ADRB1 Gly389Asp SNP reduces response to beta-blockade in subjects with permanent AF.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be at least 18 years of age.
* Subjects must have a history of persistent AF currently treated with a rate control strategy.
* Subjects should be willing to give written, informed consent.
* Subjects must be willing and able to participate in the exercise protocol.

Exclusion Criteria:

* New York Heart Association Class III or IV heart failure.
* A history of heart failure induced by tachy-arrhythmia.
* A history of coronary artery disease and the presence of at least one of the following:

  * Canadian Class III or IV angina.
  * Recent myocardial infarction, coronary artery bypass grafting, or percutaneous coronary intervention within 6 months.
* Severe renal or hepatic impairment.
* Subjects who have a clinically significant allergy/intolerance to atenolol, including a history of beta-blocker induced bronchospasm.
* Females who are pregnant or nursing.
* History of severe AV node dysfunction/pacemaker dependence.
* Subjects who have a systolic blood pressure < 90 mm Hg or resting Ventricular Rate <50 or >120 per minute on the day of the study.
* Patients currently taking Vaughan-Williams Class I or III anti-arrhythmic drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] European Heart Rhythm Association; Heart Rhythm Society; Fuster V, Ryden LE, Cannom DS, Crijns HJ, Curtis AB, Ellenbogen KA, Halperin JL, Le Heuzey JY, Kay GN, Lowe JE, Olsson SB, Prystowsky EN, Tamargo JL, Wann S, Smith SC Jr, Jacobs AK, Adams CD, Anderson JL, Antman EM, Hunt SA, Nishimura R, Ornato JP, Page RL, Riegel B, Priori SG, Blanc JJ, Budaj A, Camm AJ, Dean V, Deckers JW, Despres C, Dickstein K, Lekakis J, McGregor K, Metra M, Morais J, Osterspey A, Zamorano JL; American College of Cardiology; American Heart Association Task Force on Practice Guidelines; European Society of Cardiology Committee for Practice Guidelines; Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation. ACC/AHA/ESC 2006 guidelines for the management of patients with atrial fibrillation--executive summary: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and the European Society of Cardiology Committee for Practice Guidelines (Writing Committee to Revise the 2001 Guidelines for the Management of Patients With Atrial Fibrillation). J Am Coll Cardiol. 2006 Aug 15;48(4):854-906. doi: 10.1016/j.jacc.2006.07.009. No abstract available. PMID 16904574
- [Background] Go AS, Hylek EM, Phillips KA, Chang Y, Henault LE, Selby JV, Singer DE. Prevalence of diagnosed atrial fibrillation in adults: national implications for rhythm management and stroke prevention: the AnTicoagulation and Risk Factors in Atrial Fibrillation (ATRIA) Study. JAMA. 2001 May 9;285(18):2370-5. doi: 10.1001/jama.285.18.2370. PMID 11343485
- [Background] Miyasaka Y, Barnes ME, Gersh BJ, Cha SS, Bailey KR, Abhayaratna WP, Seward JB, Tsang TS. Secular trends in incidence of atrial fibrillation in Olmsted County, Minnesota, 1980 to 2000, and implications on the projections for future prevalence. Circulation. 2006 Jul 11;114(2):119-25. doi: 10.1161/CIRCULATIONAHA.105.595140. Epub 2006 Jul 3. PMID 16818816
- [Background] Beta-Blocker Evaluation of Survival Trial Investigators; Eichhorn EJ, Domanski MJ, Krause-Steinrauf H, Bristow MR, Lavori PW. A trial of the beta-blocker bucindolol in patients with advanced chronic heart failure. N Engl J Med. 2001 May 31;344(22):1659-67. doi: 10.1056/NEJM200105313442202. PMID 11386264
- [Background] Havlik RJ, Garrison RJ, Fabsitz R, Feinleib M. Variability of heart rate, P-R, QRS and Q-T durations in twins. J Electrocardiol. 1980;13(1):45-8. doi: 10.1016/s0022-0736(80)80008-2. PMID 7188949
- [Background] Hanson B, Tuna N, Bouchard T, Heston L, Eckert E, Lykken D, Segal N, Rich S. Genetic factors in the electrocardiogram and heart rate of twins reared apart and together. Am J Cardiol. 1989 Mar 1;63(9):606-9. doi: 10.1016/0002-9149(89)90907-7. PMID 2919564
- [Background] Levin MC, Marullo S, Muntaner O, Andersson B, Magnusson Y. The myocardium-protective Gly-49 variant of the beta 1-adrenergic receptor exhibits constitutive activity and increased desensitization and down-regulation. J Biol Chem. 2002 Aug 23;277(34):30429-35. doi: 10.1074/jbc.M200681200. Epub 2002 May 28. PMID 12034720
- [Background] Mason DA, Moore JD, Green SA, Liggett SB. A gain-of-function polymorphism in a G-protein coupling domain of the human beta1-adrenergic receptor. J Biol Chem. 1999 Apr 30;274(18):12670-4. doi: 10.1074/jbc.274.18.12670. PMID 10212248
- [Background] Sandilands A, Yeo G, Brown MJ, O'Shaughnessy KM. Functional responses of human beta1 adrenoceptors with defined haplotypes for the common 389R>G and 49S>G polymorphisms. Pharmacogenetics. 2004 Jun;14(6):343-9. doi: 10.1097/00008571-200406000-00003. PMID 15247626
- [Background] Mialet Perez J, Rathz DA, Petrashevskaya NN, Hahn HS, Wagoner LE, Schwartz A, Dorn GW, Liggett SB. Beta 1-adrenergic receptor polymorphisms confer differential function and predisposition to heart failure. Nat Med. 2003 Oct;9(10):1300-5. doi: 10.1038/nm930. Epub 2003 Sep 14. PMID 14502278
- [Background] Liu J, Liu ZQ, Yu BN, Xu FH, Mo W, Zhou G, Liu YZ, Li Q, Zhou HH. beta1-Adrenergic receptor polymorphisms influence the response to metoprolol monotherapy in patients with essential hypertension. Clin Pharmacol Ther. 2006 Jul;80(1):23-32. doi: 10.1016/j.clpt.2006.03.004. Epub 2006 Jun 8. PMID 16815314
- [Background] Johnson JA, Zineh I, Puckett BJ, McGorray SP, Yarandi HN, Pauly DF. Beta 1-adrenergic receptor polymorphisms and antihypertensive response to metoprolol. Clin Pharmacol Ther. 2003 Jul;74(1):44-52. doi: 10.1016/S0009-9236(03)00068-7. PMID 12844134
- [Background] Small KM, Forbes SL, Rahman FF, Bridges KM, Liggett SB. A four amino acid deletion polymorphism in the third intracellular loop of the human alpha 2C-adrenergic receptor confers impaired coupling to multiple effectors. J Biol Chem. 2000 Jul 28;275(30):23059-64. doi: 10.1074/jbc.M000796200. PMID 10801795
- [Background] Lobmeyer MT, Gong Y, Terra SG, Beitelshees AL, Langaee TY, Pauly DF, Schofield RS, Hamilton KK, Herbert Patterson J, Adams KF Jr, Hill JA, Aranda JM Jr, Johnson JA. Synergistic polymorphisms of beta1 and alpha2C-adrenergic receptors and the influence on left ventricular ejection fraction response to beta-blocker therapy in heart failure. Pharmacogenet Genomics. 2007 Apr;17(4):277-82. doi: 10.1097/FPC.0b013e3280105245. PMID 17496726
- [Background] Kaab S, Darbar D, van Noord C, Dupuis J, Pfeufer A, Newton-Cheh C, Schnabel R, Makino S, Sinner MF, Kannankeril PJ, Beckmann BM, Choudry S, Donahue BS, Heeringa J, Perz S, Lunetta KL, Larson MG, Levy D, MacRae CA, Ruskin JN, Wacker A, Schomig A, Wichmann HE, Steinbeck G, Meitinger T, Uitterlinden AG, Witteman JC, Roden DM, Benjamin EJ, Ellinor PT. Large scale replication and meta-analysis of variants on chromosome 4q25 associated with atrial fibrillation. Eur Heart J. 2009 Apr;30(7):813-9. doi: 10.1093/eurheartj/ehn578. Epub 2009 Jan 13. PMID 19141561

RESULTS

PARTICIPANT FLOW:
Groups:
- Atenolol: Ancestral Alleles: Patients will undergo a standardized, graded exercise protocol before and after receiving a dose of oral atenolol.
  participants have Ancestral Alleles
- Atenolol: Variant Carriers: Patients will undergo a standardized, graded exercise protocol before and after receiving a dose of oral atenolol.
  participants have Variant Carriers
Period: Overall Study
Arm/Group | Atenolol: Ancestral Alleles | Atenolol: Variant Carriers
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI of this study left Vanderbilt. Limited data are available for this study. Baseline data are not available per-arm, therefore, only the baseline data for overall population is being reported.
Groups:
- All Participants: all participants
Arm/Group | All Participants
Number analyzed (Participants) | 38
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 70.5 [60 to 74.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Pre- and Post-atenolol Ventricular Rate Response After 5 Minutes of Exercise
Description: After baseline vital signs and ECG are recorded, patients will be asked to perform a baseline standardized (modified Bruce) exercise protocol. Heart rate will be recorded during each stage of the exercise protocol. Patients will be asked to exercise to sub-maximal exertion. After the baseline exercise protocol, patients will be given a single dose of oral atenolol. After a two hour waiting period to allow for peak effect of atenolol, patients will repeat the exercise protocol. The primary study outcome measure will be the difference in pre- and post-atenolol ventricular rate response to exercise. The primary outcome measure will be compared in patients with various polymorphisms in genes that might play a role in the inter-individual response to atenolol.
Time Frame: after 5minutes of exercise
Measure: Mean (95% Confidence Interval); unit: beats per minute
Groups:
- Atenolol: Ancestral Alleles: Patients will undergo a standardized, graded exercise protocol before and after receiving a dose of oral atenolol.
  These patients have Ancestral Alleles
- Atenolol: Variant Carriers: Patients will undergo a standardized, graded exercise protocol before and after receiving a dose of oral atenolol.
  These patients have Variant Carriers
Arm/Group | Atenolol: Ancestral Alleles | Atenolol: Variant Carriers
Number analyzed (Participants) | 19 | 19
beats per minute | -10 [-18.6 to -1.4] | -13 [-20.2 to -5.8]

2. Primary Outcome: Change in Pre- and Post-atenolol Ventricular Rate Response After 10 and 15 Minutes of Exercise
Description: as for outcome 1
Time Frame: after 10 amd 15 minutes of exercise
Measure: Mean (95% Confidence Interval); unit: beats per minute
Arm/Group | Atenolol: Ancestral Alleles | Atenolol: Variant Carriers
Number analyzed (Participants) | 19 | 19
beats per minute
  After 10 minutes | -11 [-21.9 to -0.1] | -19.7 [-25.6 to -13.9]
  After 15 minutes | -25.5 [-67 to -16.8] | -35.2 [-53.3 to -17.1]

ADVERSE EVENTS:
Time Frame: during study visit, 1 day
Arm/Group | Atenolol: Ancestral Alleles | Atenolol: Variant Carriers
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes